CLINICAL TRIAL: NCT06647082
Title: Engaging Kids and Improving Rehab Outcomes by Gamification of Robotic Exoskeletons Combined With Proprioceptive Biofeedback
Brief Title: Engaging Kids With Robotic Exoskeletons and Gamification
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia Institute of Technology (Other)
Collaborators: Children's Healthcare of Atlanta (Other)
Responsible Party: Principal Investigator, Kinsey Herrin, Senior Research Scientist, Georgia Institute of Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: H24360
Record Dates: First submitted 2024-10-16; First posted 2024-10-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Genu Recurvatum; Crouch Gait
Keywords: Pediatric walking impairment; Exoskeleton; Knee exoskeleton; Knee hyperextension; Knee crouch gait

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Pediatric Knee Exoskeleton (Experimental): N=5 patient participants will undergo 5 sessions of experimental therapeutic rehabilitation sessions with the exoskeleton and the visual biofeedback game. Participants will use the device for a maximum of 2 hours per session for 5 sessions.
  Interventions: Device: Pediatric Knee Exoskeleton

INTERVENTIONS:
Device: Pediatric Knee Exoskeleton — The current knee exoskeleton is designed specifically for use in children. The device can be operated either bilaterally or unilaterally and is capable of providing 10- 17.4 Nm of torque assistance at the knee joint which is ~60% of the average biological joint torque for an American 15 year old child. It is adjustable in height such that the passive hip joint and powered knee joint can be placed at the correct anatomical location for each child. Thigh and calf cuffs are interchangeable to accommodate varying leg sizes. The device is autonomous, allowing a child to move freely and can even be used outdoors. The device can accommodate for varying lower limb alignment presentations, adjusting to accommodate for varying femoral rotations and varum and valgum alignments at the knee. The device can be worn independently of the visual biofeedback video game, but is intended for participants to use in conjunction with the knee exoskeleton.

SUMMARY:
Conduct a clinical field trial at CHOA's Day Rehab Program using the clinical exoskeleton in conjunction with visual biofeedback with pediatric patients who present with genu recurvatum or crouch gait over 5 rehabilitation visits.

DETAILED DESCRIPTION:
For children, mobility is a crucial activity of daily living and age-appropriate play, influencing their independence and overall quality of life. However, children with physical disabilities often experience participation restrictions especially related to physical activity. The ICF (International Classification of Functioning, Disability and Health) notes that participation is a key contributor toward a person's overall quality of life. However, children with disabilities often experience significant participation restrictions especially related to physical activity with some studies citing that less than half of children with disabilities are physically active. Participation in physical activity allows for all the benefits associated with social engagement, belonging and autonomy, influencing a child's independence and overall development. Additionally, physical activity provides the benefits of improved health related fitness, including strength and flexibility. For children with gait impairments, lack of independence may hinder development and then compound through further loss of mobility. Some of the most encountered pediatric pathologies (CP, Spina Bifida and TBI) impact physical mobility, and clinical presentations often present with aberrant motor control of the knee. Clinical presentations may vary between genu recurvatum or crouch gaits and can be confounded with various lower limb alignment presentations as well. These abnormal walking patterns can lead to detrimental long-term effects including increased stress on soft tissue structures which often leads to permanent joint deformity if left untreated, reduced locomotion capability/ independence, increased energy expenditure and pain. The investigator team has developed an autonomous bilateral research-grade pediatric knee exoskeleton, and the investigators' data on N=10 children show the investigators have addressed an initial need for an effective pediatric knee exoskeleton from previous work. However, work is still needed to encourage: 1. real-world accessibility and usability of the device in a clinic setting outside of the research laboratory, 2. long-term retention of the intervention beyond the immediate therapeutic session, and 3. fun and active patient engagement during exoskeleton use. In this study, the investigators aim to develop and test a clinically friendly, pediatric knee exoskeleton integrated with a visual biofeedback video game to improve gait related outcomes and contribute toward improved mobility in children with walking impairment. Early intervention to engage children in their rehab along with enjoyable participation may lead to improved long-term outcomes for children and their families.

The investigators will conduct a small-scale feasibility study in which N=5 patient participants will undergo 5 sessions of experimental therapeutic rehabilitation sessions with the exoskeleton and the visual biofeedback game. Participants will use the device for a maximum of 2 hours per session for 5 sessions. Sessions will be scheduled as is convenient for the participant's schedule with a goal of having one night and no more than 1 week between consecutive sessions. Outcomes will be monitored before and after each session.

The investigators hypothesize that patient outcomes, inclusive of both functional and patient reported metrics, will significantly improve from the initial baseline visit to the final evaluation after 5 sessions of therapy. Finally, the investigators will analyze the device efficacy and family/therapist survey data to implement improvements to the exoskeleton and biofeedback game in the future.

ELIGIBILITY:
Inclusion Criteria:

* Age 4-21 years
* Clinical presence of genu recurvatum or crouch gait during walking
* Ability to walk nonstop for at least 6 minutes
* Willing to participate in 5 sessions of therapy with the device with each session lasting no more than 2 hours

Exclusion Criteria:

* Inability to take commands from research staff
* Receipt of Botox injection during study trial will disqualify the participant from participating further
* Presence of uncontrolled seizures
* Non-English speaking

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Estimated)
Dates: Start 2026-06-30 (Estimated); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
10 meter walk test | 5 weeks
  The participant walks a 10 meter distance while their speed is recorded. Higher speeds are indicative of a more positive outcome.
2 minute walk test | 5 weeks
  The participant walks as far as they can walk in a period of 2 minutes and the distance is recorded. Greater distances are indicative of improved performance.
Modified Timed Up and Go | 5 weeks
  Participants are seated in a stable stool selected according to the height of subjects. The stool is positioned such that it does not move when the participant moves from sitting to standing. Participant is seated with feet flat on the floor in such a way that hip and knee remained in 90° of flexion. A marking tape was used to stick a star mark on the wall at a distance of 3 m from the chair. Participant is instructed to stand up, walk, touch the star and sit back down while being timed. Shorter times are indicative of improved performance.

SECONDARY OUTCOMES:
Gillette Functional Assessment Questionnaire | 5 weeks
  Family/patient reported survey which asks questions about their perception of the child's mobility.

CONTACTS AND LOCATIONS:
Overall Officials: Kinsey Herrin, MSPO, Principal Investigator — Georgia Institute of Technology
Locations (1):
- Children's Healthcare of Atlanta - Scottish Rite, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No